CLINICAL TRIAL: NCT06496100
Title: Effect of Triticum Aestivum on Appetite Regulation and the Ghrelin, Leptin, Adiponectin Hormonal Axis in Patients With Obesity
Brief Title: Effect of Triticum Aestivum on Appetite, Ghrelin, Leptin, Adiponectin Hormonal Axis in Patients With Obesity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2023-1301-251
Record Dates: First submitted 2024-03-26; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Leptin Deficiency; Ghrelin; Adiponectin
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial, of two parallel groups, double blind, with random assignment and control group.
  38 patients:
  1. 19 patients with 500 mg of triticum aestivum orally every 12 hours for 120 days.
  2. 19 patients with 500 mg of placebo orally every 12 hours for 120 days.
     * Visit 1/ Day -7: Screening period, information about the study, signing of informed consent, medical history, anthropometric measurements, baseline laboratory tests.
     * Visit 2/Day 0: Randomization, 60 tablets of Triticum aestivum or placebo will be given, general diet and exercise recommendations.
     * Visit 3,4,5/Day 30,60,90: Treatment adherence evaluation, laboratory tests, adverse events evaluation, general diet and exercise recommendations and 60 tablets of Triticum aestivum or placebo will be given.
     * Visit 6/Final/Day 120 ÷ 7: Anthropometric measurements will be taken, laboratory tests will be performed, adherence to treatment and adverse events will be
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) All participants will be submitted to the selection of a sealed envelope which will have a numerical code previously defined by a third party for each intervention group.
  The total number of envelopes required to complete the minimum number of participants will have numerical codes that identify the bottle of intervention treatment that should receive the participant during the intervention period.
  They will be divided into half blinded codes for triticum aestivum group and half for placebo to complete the size of each subsample. Chance guarantees blinding, neither the participant nor the researcher will know the type of treatment. The database for the blinded statistical analysis will be completed. The blind man will be removed once the statistical analysis has been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triticum aestivum (Active Comparator): A group of 19 patients with a diagnosis of obesity without pharmacological or surgical treatment, who will receive 500 mg of triticum aestivum orally every 12 hours for 120 days.
  Interventions: Drug: Triticum Aestivum
- Placebo (calcined magnesia) (Placebo Comparator): A group of 19 patients with a diagnosis of obesity without pharmacological or surgical treatment, who will receive 500 mg of calcined magnesia orally every 12 hours for 120 days.
  Interventions: Drug: Placebo (calcined magnesia)

INTERVENTIONS:
Drug: Triticum Aestivum — The intervention period will be 120 days, looking for effects on appetite regulation and the hormonal axis Leptin, Ghrelin and Adiponectin.
  Arms: Triticum aestivum
Drug: Placebo (calcined magnesia) — The intervention period will be 120 days, looking for effects on appetite regulation and the hormonal axis Leptin, Ghrelin and Adiponectin.
  Other Names: Calcined magnesia
  Arms: Placebo (calcined magnesia)

SUMMARY:
Obesity represents one of the major health problems worldwide; it is clear that current approaches to address obesity are largely unsuccessful. The endocrine axis of leptin and ghrelin acts as the critical link between adipose tissue and hypothalamic centers that regulate food intake, satiety, energy expenditure and weight.

Despite being a highly prevalent disease with major complications, current therapeutic options are not sufficient, as they are not ideal for the entire population. The importance of new pharmacological interventions that can be evaluated in the population at risk as an early form of treatment to avoid the development of chronic diseases with high morbidity and mortality.

Natural products such as Triticum aestivum and their high content of bioactive principles have been described for their pharmacokinetic functions in weight reduction, insulin resistance and modulation of neuropeptides involved in food intake.

DETAILED DESCRIPTION:
A double-blind clinical trial is proposed, with two parallel groups, with random assignment and group control. The universe of the sample will be patients with a diagnosis of obesity, residents of the Guadalajara Metropolitan Area, who agree to participate by signing informed consent and can go to the Biomedical Unit 02 of the Mexican Institute of Social Security.

Two parallel groups, with randomization by software using envelopes, will require a total of 38 patients, which will be distributed as follows: 1) A group of 19 patients with a diagnosis of obesity without pharmacological or surgical treatment, who will receive 500 mg capsules with lyophilized Triticum aestivum orally every 12 hours for 120 days, and 2) A group of 19 patients with a diagnosis of obesity without pharmacological or surgical treatment, who will receive 500 mg capsules of placebo (calcined magnesia) orally every 12 hours for 120 days.

ELIGIBILITY:
Inclusion Criteria:

People of any sex (eumenorrheic women with mechanical or definitive contraceptive method without hormonal treatment).

Age from 30 to 50 years old. Residents of the metropolitan area of Guadalajara. Signed informed consent form. People with a diagnosis of obesity (BMI ≥30 - 39.9 kg/m2), stable body weight within the 3 months prior to the start of the study.

Exclusion Criteria:

Diagnosis of diabetes and dyslipidemia. Diagnosis of anxiety and/or depression. History of: liver disease, chronic kidney disease, thyroid disease, cancer. Antidiabetic treatment, lipid-lowering, food supplements, antidepressants, corticosteroids.

Acute infectious processes Alcoholism and/or active smoking in any intensity within the 12 months prior to the start of the study.

Suspected or confirmed pregnancy or breastfeeding. History of drug intake. Recent surgery (<3 months) Carrying a pacemaker, or any other bioelectronic or metallic element. Excessive sedentary lifestyle defined as physical activity less than the equivalent of 15 minutes of walking per day.

Excessive exercise, defined as physical activity equivalent to running for 60 minutes per day.

Intake of anorexigenic drugs, hypolipidemic drugs or drugs with effect on body weight.

History of any type of cancer, hyperthyroidism, hypothyroidism, renal disease, liver disease and pancreatic disease.

History of hypersensitivity to the study drug (gluten).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-11-27 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of Triticum aestivum on leptin in patients with obesity. | 120 days
  To quantify the serum concentrations of leptin ( pg/mL) before and after of treatment with 1000 mg of Triticum aestivum or placebo.
To evaluate the effect of Triticum aestivum on ghrelin in patients with obesity. | 120 days
  To quantify the serum concentrations of ghrelin ( pg/mL) before and after of treatment with 1000 mg of Triticum aestivum or placebo.
To evaluate the effect of Triticum aestivum on adiponectin in patients with obesity. | 120 days
  To quantify the serum concentrations of adiponectin ( pg/mL) before and after of treatment with 1000 mg of Triticum aestivum or placebo.
To evaluate the effect of Triticum aestivum on satiety regulation | 120 days
  To evaluate the effect on satiety by the visual analog scale for satiety and appetite
To evaluate the effect of Triticum aestivum on appetite regulation | 120 days
  To evaluate the effect on satiety by the visual analog scale for satiety and appetite

CONTACTS AND LOCATIONS:
Overall Officials: Sandra O Hernandez Gonzalez, PhD, Principal Investigator — Instituto Mexicano del Seguro Social, Unidad de Investigación Biomédica 02
Locations (1):
- Biomedical Unit Research 02, Specialties Hospital, Medical Unit of High Specialty, West National Medical Center, Mexican Social Security Institute., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All data resulting from the clinical investigation, except the personal identification of the subjects (name, address, telephone, etc.)
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication.
Access Criteria: The data can be shared through a request addressed to the principal investigator Dr. Sandra Ofelia Hernández González, basing the reason for what they are requested

REFERENCES:
- See also: Hypothalamic IKKβ/NF-κB and ER Stress Link Overnutrition to Energy Imbalance and Obesity. — http://linkinghub.elsevier.com/retrieve/pii/S0092867408010088
- See also: Issues in Measuring and Interpreting Human Appetite (Satiety/Satiation) and Its Contribution to Obesity. — http://link.springer.com/10.1007/s13679-019-00340-6
- See also: Eating and Weight Disorders - Studies on Anorexia, Bulimia and Obesity — http://link.springer.com/10.1007/s40519-013-0094-z
- See also: Proanthocyanidins potentiate hypothalamic leptin/STAT3 signalling and Pomc gene expression in rats with diet-induced obesity. — http://www.nature.com/articles/ijo2016169
- See also: Active ingredients from natural botanicals in the treatment of obesity. — http://onlinelibrary.wiley.com/doi/10.1111/obr.12228
- See also: Hunger and Satiety Mechanisms and Their Potential Exploitation in the Regulation of Food Intake. — http://link.springer.com/10.1007/s13679-015-0184-5
- See also: STAT3 signalling is required for leptin regulation of energy balance but not reproduction. — http://www.nature.com/articles/nature01388
- See also: Microglia Dictate the Impact of Saturated Fat Consumption on Hypothalamic Inflammation and Neuronal Function. — http://linkinghub.elsevier.com/retrieve/pii/S2211124714009723
- See also: Leptin and the Regulation of Body Weigh. — http://www.jstage.jst.go.jp/article/kjm/60/1/60_1_1/_article
- See also: Positional cloning of the mouse obese gene and its human homologue. — http://www.nature.com/articles/372425a0
- See also: The cellular and molecular bases of leptin and ghrelin resistance in obesity. — http://www.nature.com/articles/nrendo.2016.222
- See also: Integrative physiology of human adipose tissue. — http://www.nature.com/articles/0802326
- See also: Regulation of Jak Kinases by Intracellular Leptin Receptor Sequences. — http://linkinghub.elsevier.com/retrieve/pii/S0021925819719954